CLINICAL TRIAL: NCT04022395
Title: Concordance Between Stress CMR and Coronary Angiography in Pediatric Patients With Suspected Coronary Artery Disease
Brief Title: Stress CMR in Pediatric Patients With Suspected Coronary Artery Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Istituto Giannina Gaslini (Other)
Responsible Party: Principal Investigator, Nicola Stagnaro, MD, Principal Investigator, Radiology Dept, Cardiovascular MRI Team, Istituto Giannina Gaslini
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 519REG2016
Record Dates: First submitted 2019-03-15; First posted 2019-07-17 (Actual); Last update posted 2021-09-08 (Actual); Status verified 2021-09

CONDITIONS: Coronary Disease
MeSH Terms: conditions — Coronary Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- stress cardiac MRI (Experimental): * To optimize the scan protocol and the sequence parameters
  * To investigate the clinical compliance of stress induced cardiac MRI in pediatric patients
  * To test the ability of stress cMRI to visualize coronary arteries morphological irregularities, the corresponding wall motion abnormalities and perfusion - viability features
  Interventions: Diagnostic Test: stress cardiac MRI

INTERVENTIONS:
Diagnostic Test: stress cardiac MRI — pharmacological stress testing has evolved as an alternative to physical exercise for the detection of inducible myocardial ischemia

SUMMARY:
stress cMRI with Dobutamine stress agent (stress cMRI), represent the combination of two orders of exams routinely performed (cMRI and stress diagnostic series of exams) without additional risk for the patient, but with the advantage of non-invasiveness and lack of radiation, and less laborious for the participants

DETAILED DESCRIPTION:
Surgical revascularization or angioplasty are therapeutic options for coronary lesions even in infants and children. Pharmacological stress induced cMRI could provide crucial information such as coronary arteries origin and proximal pathway, wall motion abnormalities, myocardial perfusion and viability, enabling accurate monitoring of symptomatic and non-pediatric patients. Investigators would build a prospective series of stress cMRI exams in pediatric symptomatic and non-patients, with suspected or previously diagnosed coronary artery disease. Investigators would put the results in comparison with ECG, Exercise test, stress Cardiac Ultrasound and Angiography. At the end of the study, if supported by results, the aim is to replace the current diagnostic procedure (ECG, Exercise test, stress Cardiac Ultrasound and Angiography) which need long hospitalization, expose the patient to radiation dose, is uncomfortable for the patient, and is characterized by a non-negligible risk due to invasive procedure, with a single exam (stress cMRI) which is dose-free, minimal risk related, without hospitalization, and less expensive for National Care System.

ELIGIBILITY:
Inclusion Criteria:

* Between 8 and 18 years-old patients symptomatic and non, with suspected or previously diagnosed coronary arteries disease

  * Coronary artery re-implantation after arterial switch
  * ALCAPA Syndrome, and other anomalies of origin or pathway
  * replacement of aortica valve with pulmonary autograft (Ross procedure)
  * Kawasaki disease
  * primary dilatative cardiomyopathy
  * coronary atresia
  * familiar Hypercholesterolemia
  * bicuspid aortic valve
  * chest pain
  * exertional dyspnea of suspected coronary artery nature
  * coronary artery fistula

Exclusion Criteria:

* General contraindication to MRI (non MRI compatible device: vascular clips, foreign bodies, coronary and peripheral artery stents, aortic stent grafts, prosthetic heart valves and annuloplasty rings, cardiac occluder devices, vena cava filters and embolisation coils, haemodynamic monitoring and temporary pacing devices, haemodynamic support devices, permanent cardiac pacemakers and implantable cardioverter-defibrillators, retained transvenous pacemaker and defibrillator leads, cochlear implants, claustrophobia, pregnancy and postpartum),

  * contraindication to contrast agent (renal insufficiency, hypersensitivity to the Dotarem active substance or to any of the excipients:)
  * contraindication to stress agent (hypersensitivity to Dobutamine active substance or to any of the excipients)
  * severe arterial hypertension (>/= 220/120 mmHg)
  * unstable angina pectoris
  * significant aortic stenosis
  * complex cardiac arrhythmias including uncontrolled atrial fibrillation
  * hypertrophic obstructive cardiomyopathy
  * myocarditis, endocerditis
  * pericarditis
  * uncontrolled congestive heart failure
  * previous manifestations of hypersensitivity to dobutamine
  * refuse to join the protocol and relative off-label procedures

Ages: 8 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 15 (Actual)
Dates: Start 2018-10-18 (Actual); Primary Completion 2021-02-28 (Actual); Study Completion 2021-03-30 (Actual)

PRIMARY OUTCOMES:
Multiparameters diagnostic concordance | 24 month
  • Agreement of results between stress cMRI and the current practice constituted by Exercise test, Stress Cardiac Ultrasound and Invasive Angiography

SECONDARY OUTCOMES:
Efficacy of stress cMRI | 24 month
  Predictive value of stress cMRI to determine the incidence of post-surgical complication of switch repair, and other pathological conditions affecting coronary arteries in natural history, in comparison with tradition test. This will be measured the number coronary segments affected, and consequences on wall motion abnormalities
Incidence of Treatment-Emergent Adverse Events | 24 month
  Number of participants with treatment-related adverse events as assessed by CTCAE v4.0

CONTACTS AND LOCATIONS:
Locations (1):
- Istituto Giannina Gaslini, Genova, Italy

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Study Protocol (2017-07-09): https://cdn.clinicaltrials.gov/large-docs/95/NCT04022395/Prot_001.pdf